CLINICAL TRIAL: NCT00789919
Title: Mild Preeclampsia Near Term: Deliver or Deliberate?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001-1114
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2008-11

CONDITIONS: Preeclampsia
Keywords: Mild Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Study participants (those diagnosed with mild preeclampsia) are admitted to hospital for standard inpatient management of their disease.
- 2 (Experimental): Study participants (those diagnosed with mild preeclampsia) are admitted to hospital and their infant is delivered as soon as possible after 34 weeks gestation. As there is no determined optimal time of delivery in these patients, delivery is the intervention.
  Interventions: Procedure: Delivery of infant

INTERVENTIONS:
Procedure: Delivery of infant — Vaginal delivery or cesarean section, whichever is indicated
  Arms: 2

SUMMARY:
Preeclampsia with new-onset hypertension and proteinuria is a pregnancy-specific disease that affects 5-7% of gestations usually after the 20th week. Most cases are mild, but severe cases exhibit multiple abnormalities in blood and maternal organ systems. Severe forms of preeclampsia/eclampsia are a major contributor to maternal death in the world. Delivery stops disease progression and recovery can begin. Patients with mild preeclampsia between 34-38 weeks' gestation usually are hospitalized for evaluation and close monitoring of signs, symptoms, and certain laboratory studies as reflectors of disease status. As inpatients mothers are monitored frequently for evidence of maternal or fetal compromise until 38 weeks gestation when delivery is accomplished. If a patient with mild preeclampsia labors after 34 weeks, no attempt is made to stop labor and delivery is undertaken. It remains unclear when during the third trimester that delivery should be accomplished for maximal maternal safety and minimal fetal risk. In this research project, we will identify patients who are at least 34 weeks pregnant with mild preeclampsia. After informed consent to participate in the trial, we will randomize participants to either be delivered immediately or treated with observation and maternal-fetal surveillance in hospital as described previously with delivery at 38 weeks. There will be 110 participants enrolled in each arm of the study for a total of 220 patients who will be managed in the Wiser Hospital. We intend to analyze a number of maternal and fetal outcomes including cost comparisons for the care of both mother and fetus in the two groups of randomized patients. The findings should impact care of the pregnant patient with mild preeclampsia in the third trimester with regard to how early and how late in gestation that delivery should be accomplished for optimal maternal and perinatal benefit.

ELIGIBILITY:
Inclusion Criteria:

* Mild Preeclampsia equal to or greater than 34 weeks' and less that 38 weeks' gestation singleton gestation no maternal or fetal contraindications to conservative management

Exclusion Criteria:

* Non-gestational diabetes Chronic hypertension Severe preeclampsia Non-reassuring fetal assessment intrauterine growth restriction fetal anomalies multiple gestation premature preterm rupture of membranes placenta previa unexplained vaginal bleeding antihypertensive use current gestation poor dating criteria contraindication to conservative management active labor at admission

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2002-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Progression to severe preeclampsia in the control group necessitating delivery of the infant. | End of study

SECONDARY OUTCOMES:
Maternal morbidity | End of study
Fetal morbidity and mortality | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Y Owens, M.D., Principal Investigator — University of Mississippi Medical Center
Locations (1):
- Winfred L Wiser Hospital for Women and Infants, Jackson, Mississippi, United States